CLINICAL TRIAL: NCT03044964
Title: Effect of Ranolazine on Activity Level in Patients With Angina After FFR Based Deferred Intervention
Brief Title: Effect of Ranolazine on Activity Level in Patients With Angina After FFR Based Deferred Intervention (REPTAR)
Acronym: REPTAR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amit Malhotra, MD (Industry)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, Amit Malhotra, MD, Sponsor-Investigator, Stern Cardiovascular Foundation, Inc.
Organization: Stern Cardiovascular Foundation, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REPTAR
Record Dates: First submitted 2017-01-26; First posted 2017-02-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Angina
Keywords: Angina, Chest Pain
MeSH Terms: conditions — Angina Pectoris; Chest Pain | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranolazine (Active Comparator): At randomization, patients will be started on 500mg of Ranolazine, twice daily for 1 week. After 1 week, the dosage may be increased to 1000mg of Ranolazine, twice daily for 5 weeks.
  Interventions: Drug: Ranolazine
- Placebo (Placebo Comparator): At Randomization, patients will be started on 500mg of a placebo, twice daily for 1 week. After 1 week, the dosage of the placebo may be increased to 1000mg, twice daily for 5 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — Patients will be started on 500mg twice daily and may be increased to 1000mg twice daily after 1 week. Patients will or may remain on the 1000mg for 5 weeks.
  Other Names: Ranexa
  Arms: Ranolazine
Drug: Placebo — Patients will be started on 500mg twice daily and may be increased to 1000mg twice daily after 1 week. Patients will or may remain on the 1000mg for 5 weeks.
  Arms: Placebo

SUMMARY:
The post-marketing study is designed to evaluate the activity level and exercise tolerance of patients with deferred percutaneous intervention due to FFR (fractional flow reserve) greater or equal to 0.81 and treatment with Ranolazine versus placebo.

DETAILED DESCRIPTION:
Ranolazine was approved as Ranexa in the United States on January 31, 2006 for the treatment of chronic angina. This post-marketing study is a single-center, double-blind, prospective, randomized, parallel-group evaluation of patients randomized 1:1 between Ranolazine and placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be willing and able to comply with schedules visits, treatment plan, and other study procedures.
2. There must be evidence of personally signed and dated informed consent documents.
3. Subjects must have a documented history of anginal chest pain equal to or greater than one (1) episode per week prior to cardiac catheterization.
4. Subjects must have greater than or equal to one (1) episode of angina chest pain between screening visit and randomization visit.
5. Subject must have documented cardiac catheterization with deferred percutaneous intervention and fractional flow reserve (FFR) greater than or equal to 0.81 within thirty (30) days, or an (FFR) less than 0.81if not a candidate for revascularization based upon operator discretion.

   -

Exclusion Criteria:

1. Subjects with a congenital or acquired QT interval prolongation (greater than or equal to 440ms in men/greater than or equal to 460ms in women).
2. Subjects prescibed strong CYP3A inhibitors (including ketaconazole, itraconazole, clarithromycin, nefazodone, nelfinavir, ritonavir, indinavir and saquinavir.) and/or strong CYP3A inducers (rifampin, rifabutin, rifapentin, Phenobarbital, phenytoin, carbamezepine and St. John's wort).
3. Subjects prescribed to Simvastatin (Zocor) that cannot have dose reduced to appropriate levels (20mg QD) per physician or have medication discontinued during the clinical trial.
4. Subjects prescribed Metformin that cannot have dose reduced to appropriate levels (less than or equal to 850mg BID) per physician or have medication discontinued during the clinical trial.
5. Subjects prescribed Digoxin that cannot have dose reduced to appropriate levels (0.125mg QD) per physician or have medication discontinued during the clinical trial.
6. Subjects with life expectancy less than the duration of the trial.
7. Subjects with a history of liver cirrhosis.
8. Subject with chronic renal disease with creatinine clearance of less than 30mL/min.
9. Subjects participating in any other clinical trial for the duration of the trial.
10. Females who are of childbearing potential, who are unwilling or unable to use highly effective method of contraception -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01-10 (Actual); Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Within-patient comparison of accelerometer-assessed physical activity utilizing the Actigraph accelerpmeter from baseline to end of study between Ranolazine and placebo. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Amit Malhotra, MD, Principal Investigator — Stern Cardiovascular Foundation, Inc.
Locations (1):
- Stern Cardiovascular Foundation, Inc, Southaven, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belardinelli L, et al. Eur Heart J. 2004;6(suppl I):I3-I7.
- [Background] Hasenfuss G, Maier LS. Mechanism of action of the new anti-ischemia drug ranolazine. Clin Res Cardiol. 2008 Apr;97(4):222-6. doi: 10.1007/s00392-007-0612-y. Epub 2007 Nov 28. PMID 18046526
- [Background] Wagner S, Seidler T, Picht E, Maier LS, Kazanski V, Teucher N, Schillinger W, Pieske B, Isenberg G, Hasenfuss G, Kogler H. Na(+)-Ca(2+) exchanger overexpression predisposes to reactive oxygen species-induced injury. Cardiovasc Res. 2003 Nov 1;60(2):404-12. doi: 10.1016/j.cardiores.2003.08.006. PMID 14613870
- [Background] Moss AJ, Zareba W, Schwarz KQ, Rosero S, McNitt S, Robinson JL. Ranolazine shortens repolarization in patients with sustained inward sodium current due to type-3 long-QT syndrome. J Cardiovasc Electrophysiol. 2008 Dec;19(12):1289-93. doi: 10.1111/j.1540-8167.2008.01246.x. Epub 2008 Jul 25. PMID 18662191
- [Background] Javitz HS, Ward MM, Watson JB, Jaana M. Cost of illness of chronic angina. Am J Manag Care. 2004 Oct;10(11 Suppl):S358-69. PMID 15603245
- [Background] Fihn SD, Gardin JM, Abrams J, Berra K, Blankenship JC, Dallas AP, Douglas PS, Foody JM, Gerber TC, Hinderliter AL, King SB 3rd, Kligfield PD, Krumholz HM, Kwong RY, Lim MJ, Linderbaum JA, Mack MJ, Munger MA, Prager RL, Sabik JF, Shaw LJ, Sikkema JD, Smith CR Jr, Smith SC Jr, Spertus JA, Williams SV, Anderson JL; American College of Cardiology Foundation/American Heart Association Task Force. 2012 ACCF/AHA/ACP/AATS/PCNA/SCAI/STS guideline for the diagnosis and management of patients with stable ischemic heart disease: a report of the American College of Cardiology Foundation/American Heart Association task force on practice guidelines, and the American College of Physicians, American Association for Thoracic Surgery, Preventive Cardiovascular Nurses Association, Society for Cardiovascular Angiography and Interventions, and Society of Thoracic Surgeons. Circulation. 2012 Dec 18;126(25):e354-471. doi: 10.1161/CIR.0b013e318277d6a0. Epub 2012 Nov 19. No abstract available. PMID 23166211
- [Background] Serruys PW, Unger F, Sousa JE, Jatene A, Bonnier HJ, Schonberger JP, Buller N, Bonser R, van den Brand MJ, van Herwerden LA, Morel MA, van Hout BA; Arterial Revascularization Therapies Study Group. Comparison of coronary-artery bypass surgery and stenting for the treatment of multivessel disease. N Engl J Med. 2001 Apr 12;344(15):1117-24. doi: 10.1056/NEJM200104123441502. PMID 11297702
- [Background] Boden WE, O'Rourke RA, Teo KK, Hartigan PM, Maron DJ, Kostuk WJ, Knudtson M, Dada M, Casperson P, Harris CL, Chaitman BR, Shaw L, Gosselin G, Nawaz S, Title LM, Gau G, Blaustein AS, Booth DC, Bates ER, Spertus JA, Berman DS, Mancini GB, Weintraub WS; COURAGE Trial Research Group. Optimal medical therapy with or without PCI for stable coronary disease. N Engl J Med. 2007 Apr 12;356(15):1503-16. doi: 10.1056/NEJMoa070829. Epub 2007 Mar 26. PMID 17387127
- [Background] Cohen DJ, Van Hout B, Serruys PW, Mohr FW, Macaya C, den Heijer P, Vrakking MM, Wang K, Mahoney EM, Audi S, Leadley K, Dawkins KD, Kappetein AP; Synergy between PCI with Taxus and Cardiac Surgery Investigators. Quality of life after PCI with drug-eluting stents or coronary-artery bypass surgery. N Engl J Med. 2011 Mar 17;364(11):1016-26. doi: 10.1056/NEJMoa1001508. PMID 21410370
- [Background] Dagenais GR, Lu J, Faxon DP, Kent K, Lago RM, Lezama C, Hueb W, Weiss M, Slater J, Frye RL; Bypass Angioplasty Revascularization Investigation 2 Diabetes (BARI 2D) Study Group. Effects of optimal medical treatment with or without coronary revascularization on angina and subsequent revascularizations in patients with type 2 diabetes mellitus and stable ischemic heart disease. Circulation. 2011 Apr 12;123(14):1492-500. doi: 10.1161/CIRCULATIONAHA.110.978247. Epub 2011 Mar 28. PMID 21444887
- [Background] Holubkov R, Laskey WK, Haviland A, Slater JC, Bourassa MG, Vlachos HA, Cohen HA, Williams DO, Kelsey SF, Detre KM; NHLBI Dynamic Registry. Registry Investigators. Angina 1 year after percutaneous coronary intervention: a report from the NHLBI Dynamic Registry. Am Heart J. 2002 Nov;144(5):826-33. doi: 10.1067/mhj.2002.125505. PMID 12422151
- [Background] Stone PH, Gratsiansky NA, Blokhin A, Huang IZ, Meng L; ERICA Investigators. Antianginal efficacy of ranolazine when added to treatment with amlodipine: the ERICA (Efficacy of Ranolazine in Chronic Angina) trial. J Am Coll Cardiol. 2006 Aug 1;48(3):566-75. doi: 10.1016/j.jacc.2006.05.044. Epub 2006 Jun 15. PMID 16875985
- [Background] Chaitman BR, Skettino SL, Parker JO, Hanley P, Meluzin J, Kuch J, Pepine CJ, Wang W, Nelson JJ, Hebert DA, Wolff AA; MARISA Investigators. Anti-ischemic effects and long-term survival during ranolazine monotherapy in patients with chronic severe angina. J Am Coll Cardiol. 2004 Apr 21;43(8):1375-82. doi: 10.1016/j.jacc.2003.11.045. PMID 15093870
- [Background] Chestnut LG, Keller LR, Lambert WE, Rowe RD. Measuring heart patients' willingness to pay for changes in angina symptoms. Med Decis Making. 1996 Jan-Mar;16(1):65-77. doi: 10.1177/0272989X9601600115. PMID 8717601
- [Background] Tonino PA, De Bruyne B, Pijls NH, Siebert U, Ikeno F, van' t Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, Fearon WF; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention. N Engl J Med. 2009 Jan 15;360(3):213-24. doi: 10.1056/NEJMoa0807611. PMID 19144937
- [Background] DeBruyne B, et al. N Eng J Med. 2014;371:1208-1217.